CLINICAL TRIAL: NCT05284357
Title: Post Market Clinical Follow-up Study for Arthroplasty Shoulder System of FX Solutions at the Long Term Retro-Prospective, Non-Randomized, Non-Interventional Study
Brief Title: Post Market Clinical Follow-up Study for Arthroplasty Shoulder System of FX Solutions at the Long Term
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: FX Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: FX_PROTOC_CL_21-02
Record Dates: First submitted 2022-02-23; First posted 2022-03-17 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Shoulder Disease; Shoulder Fractures; Shoulder Arthroplasty for Revision of Previous Treatment
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (8):
- Group 1: Subjects implanted with HUMELOCK I & II® Anatomic Shoulder System: The number of patients implanted was defined by comparing sales' database of FX Solutions.
  97 patients were identified who could be included in this cohort in 11 investigational centers.
  subjects implanted in 2011 to 2013
  Interventions: Device: Shoulder Arthroplasty Surgery with HUMELOCK I & II® Anatomic Shoulder System
- Group 2: Subjects implanted with HUMELOCK II® Reversible System: The number of patients implanted was defined by comparing sales' database of FX Solutions.
  Number of patient to be determined following patients files in 4 investigational centers.
  subjects implanted in 2011 to 2013
  Interventions: Device: Shoulder Arthroplasty Surgery with HUMELOCK II® Reversible System
- Group 3: Subjects implanted with HUMELOCK Reversed® Shoulder System: The number of patients implanted was defined by comparing sales' database of FX Solutions.
  154 patients were identified who could be included in this cohort in 5 investigational centers.
  subjects implanted in 2012 and 2013
  Interventions: Device: Shoulder Arthroplasty Surgery with HUMELOCK Reversed® Shoulder System
- Group 4: Subjects implanted with EASYTECH® Anatomic Shoulder System: The number of patients implanted was defined by comparing sales' database of FX Solutions.
  66 patients were identified who could be included in this cohort in 5 investigational centers subjects implanted in 2013 and 2014
  Interventions: Device: Shoulder Arthroplasty Surgery with EASYTECH® Anatomic Shoulder System
- Group 5: Subjects implanted with EASYTECH® Reversed System (Primary intention): The number of patients implanted was defined by comparing sales' database of FX Solutions.
  7 patients were identified who could be included in this cohort in 5 investigational centers subjects implanted in 2013 and 2014
  Interventions: Device: Shoulder Arthroplasty Surgery with EASYTECH® Reversed System (Primary intention)
- Group 6:Subjects implanted with EASYTECH® Reversible System (Revision of Easytech Anatomic): The number of patients implanted was defined by comparing sales' database of FX Solutions.
  the number of subjects will depend of revised subjects primary implanted with Easytech Anatomic® along the dedicated period subjects implanted in 2013 to 2014
  Interventions: Device: Shoulder Arthroplasty Surgery with EASYTECH® Reversible System (for revision only)
- Group 7: Subjects implanted with HUMERIS® Anatomic Shoulder System: The number of patients implanted was defined by comparing sales' database of FX Solutions.
  11 patients were identified who could be included in this cohort in 3 investigational centers Subjects implanted in 2014 to 2015
  Interventions: Device: Shoulder Arthroplasty Surgery with HUMERIS® Anatomic Shoulder System
- Group 8: Subjects implanted with HUMERIS® Reversible Shoulder System: The number of patients implanted was defined by comparing sales' database of FX Solutions.
  72 patients were identified who could be included in this cohort in 2 investigational centers Subjects implanted in 2014 to 2015
  Interventions: Device: Shoulder Arthroplasty Surgery with HUMERIS® Reversible Shoulder System

INTERVENTIONS:
Device: Shoulder Arthroplasty Surgery with HUMELOCK I & II® Anatomic Shoulder System — HUMELOCK II® is a new-generation of modular implant designed for the effective treatment of 3 or 4 part fractures of proximal humerus. The range of cases in which it can be used is wider than a simple reconstructive anatomical prosthesis. In fact, thanks to its anchoring plate, and if cephalic perfusion criteria are met, the modular nature of HUMELOCK II® means it is possible to retain the patient's native humeral head, even in cases of severe osteopenia.
  The HUMELOCK II® shoulder prosthesis allows the reconstruction of the shoulder joint as a result of a trauma (complex fracture of the proximal humerus, a common occurrence in severely injured shoulders. The HUMELOCK II® shoulder system may also be suitable for treating cases of failure of an existing shoulder prosthesis where a stem or other locking mechanism may be needed. The HUMELOCK II® shoulder prosthesis is a hemi shoulder and a total shoulder prosthesis.
  Groups: Group 1: Subjects implanted with HUMELOCK I & II® Anatomic Shoulder System
Device: Shoulder Arthroplasty Surgery with HUMELOCK II® Reversible System — HUMELOCK II® is a new-generation of modular implant designed for the effective treatment of 3 or 4 part fractures of proximal humerus.
  The HUMELOCK II® shoulder prosthesis allows the reconstruction of the shoulder joint as a result of a trauma (complex fracture of the proximal humerus). It is designed for use in complex shoulder reconstruction procedures in patients with stage 3 or 4 fragments in the proximal humerus - a common occurrence in severely injured shoulders. The HUMELOCK II® reversible system may also be suitable for treating cases of failure of an existing shoulder prosthesis where a stem or other locking mechanism may be needed.
  The HUMELOCK II reversible system is used when the rotator cuff is injured.
  Groups: Group 2: Subjects implanted with HUMELOCK II® Reversible System
Device: Shoulder Arthroplasty Surgery with HUMELOCK Reversed® Shoulder System — Humelock Reversed® is a new generation of reversed prosthesis, designed for numerous shoulder pathologies: ranging from offset arthritis to a complex cephalotuberosity fracture. A centric or eccentric glenosphere, tilted at 10°, centered on a variable length baseplate post and the position of which is guided by an intuitive adaptive instrumentation. A 145° prosthetic epiphysis allows the pillar of the scapula to be protected while maintaining optimum stability. The humeral implant is positioned naturally in the center of the epiphysis, preserving the remaining bone as much as possible. Options of locking or cementing will allow the surgeon to position the prosthetic stem at the required height, according to the patient's indication and anatomy. The surgery is called total shoulder arthroplasty. It is also indicated in a failed hemi-arthroplasty or a failed total arthroplasty. It is indicated for significant rupture of rotator cuff-tear (first surgery or revision surgery)
  Groups: Group 3: Subjects implanted with HUMELOCK Reversed® Shoulder System
Device: Shoulder Arthroplasty Surgery with EASYTECH® Anatomic Shoulder System — EASYTECH Anatomical Shoulder System is indicated for use in total shoulder replacement to treat a severely painful and/or disabled joint resulting from osteoarthritis or rheumatoid arthritis.
  EASYTECH system is a new generation of modular implant designed for the reconstruction of the shoulder joint for treating cases of degenerative pathology. The surgery is called total shoulder arthroplasty. EASYTECH prosthesis is a stemless system of shoulder components. It is a bone-preserving implant. The anchor base provides primary stability to pulling-out thanks to peripheral pegs in the shape of fir trees and their asymmetric orientations ensure its rotational stability
  Groups: Group 4: Subjects implanted with EASYTECH® Anatomic Shoulder System
Device: Shoulder Arthroplasty Surgery with EASYTECH® Reversed System (Primary intention) — EASYTECH Reversed Shoulder System is indicated for primary total shoulder arthroplasty for the relief of pain and to improve function in patients with a massive and non-repairable rotator cuff tear.
  EASYTECH system is a new generation of modular implant designed for the reconstruction of the shoulder joint for treating cases of degenerative pathology. . EASYTECH prosthesis is a stemless system of shoulder components. It is a bone-preserving implant. The anchor base provides primary stability to pulling-out thanks to peripheral pegs in the shape of fir trees and their asymmetric orientations ensure its rotational stability. A centric or eccentric glenosphere, tilted at 10°, centered on a variable length baseplate post (compatible with positioning techniques), and the position of which is guided by an intuitive adaptive instrumentation
  Groups: Group 5: Subjects implanted with EASYTECH® Reversed System (Primary intention)
Device: Shoulder Arthroplasty Surgery with EASYTECH® Reversible System (for revision only) — EASYTECH Reversible Shoulder System is indicated for revision total shoulder arthroplasty for the relief of pain and to improve function in patients with a massive and non-repairable rotator cuff tear.
  EASYTECH system is a new generation of modular implant designed for the reconstruction of the shoulder joint for treating cases of degenerative pathology. . EASYTECH prosthesis is a stemless system of shoulder components. It is a bone-preserving implant. The anchor base provides primary stability to pulling-out thanks to peripheral pegs in the shape of fir trees and their asymmetric orientations ensure its rotational stability. A centric or eccentric glenosphere, tilted at 10°, centered on a variable length baseplate post (compatible with positioning techniques), and the position of which is guided by an intuitive adaptive instrumentation.
  Groups: Group 6:Subjects implanted with EASYTECH® Reversible System (Revision of Easytech Anatomic)
Device: Shoulder Arthroplasty Surgery with HUMERIS® Anatomic Shoulder System — The HUMERIS Shoulder system is intended to be used in adult patients with glenohumeral joint degenerative pathologies associated or not with rotator cuff arthropathy or tears when all other non-invasive treatments have failed to reduce the pain or improve the quality of life. The HUMERIS shoulder is a system of short stem.The technical characteristics of this implant have been designed based on computer simulations, correlated to results previously published in medical journals. A 145° prosthetic epiphysis allows the pillar of the scapula to be protected while maintaining optimum stability. The humeral implant is positioned naturally in the center of the epiphysis, preserving the remaining bone as much as possible.
  Groups: Group 7: Subjects implanted with HUMERIS® Anatomic Shoulder System
Device: Shoulder Arthroplasty Surgery with HUMERIS® Reversible Shoulder System — The HUMERIS Shoulder system is intended to be used in adult patients with glenohumeral joint degenerative pathologies associated or not with rotator cuff arthropathy or tears when all other non-invasive treatments have failed to reduce the pain or improve the quality of life. The HUMERIS shoulder is a system of short stem.The technical characteristics of this implant have been designed based on computer simulations, correlated to results previously published in medical journals, in order to avoid the disadvantages of traditional reverse prostheses. A centric or eccentric glenosphere, tilted at 10°, centered on a variable length baseplate post, the position of which is guided by an intuitive adaptive instrumentation.A 145° prosthetic epiphysis allows the pillar of the scapula to be protected while maintaining optimum stability.The humeral implant is positioned naturally in the center of the epiphysis, preserving the remaining bone as much as possible
  Groups: Group 8: Subjects implanted with HUMERIS® Reversible Shoulder System

SUMMARY:
This study takes place in the framework of the Post-Market Clinical Follow-up of the FX Solutions Shoulder System. The goal of this PMCF study is to collect clinical data in order to confirm the safety and the performance at a long term and mainly the first two years of sales for each studied ranges.

Eligible patients who received the FX Solutions Shoulder System and are at about 7 years post-operative were contacted by the Investigator to explain the study, the retrospective collection and the prospective follow-up visit. Investigator also explain the analysis of the post-operative outcomes of the patient. During the call of the investigator, the patient was informed about the study's goal and about the data collection. The oral agreement of the patient was checked by the investigators in CRF with its signature. Then, an information form explaining the purpose of the data collection was provided to the patient by postmail.

The retrospective data were collected in a paper CRF via the medical file of patient.

Post-operative follow-up for all patients is limited to a teleconsultation intended to assess the patient's current condition and clinical outcomes.

Patient who are enrolled in the study shall be assigned a unique Subject Identification Number to de-identify their information.

DETAILED DESCRIPTION:
Inclusion Criteria

* Adult patient (≥ 18 years old) who received one of FX Solutions Shoulder System for indication of hemi or total shoulder replacement.
* Patient implanted between 2011 and 2015 with a minimum follow-up of 7 years
* Patient has been informed of his participation in a clinical study and did not object to data collection
* Patient insured with a social security system

Exclusion Criteria

* Patient who does not meet the inclusion criteria above
* Protected adult
* People deprived of their liberty

Study Objectives

* Primary Objective: To assess functional improvement according to the Constant score evolution compared to its preoperative value
* Secondary Objectives, assessment of:

To assess against the preoperative value:

* the Subjective Shoulder Value score evolution
* the American Shoulder and Elbow Surgeons shoulder score evolution To describe in real life
* The complications rate
* The long-term range of motion
* The revision rates and the prosthesis survival curve

Endpoints

* Primary Endpoint will be the current Constant score (measured during the assessment). The functional improvement will be evaluated according to the evolution of this score compared to its preoperative value.
* Secondary Endpoints:

Current ASES and SSV scores Current range of Motion Revision rate at a long-term follow-up. Calculation of the survival rates The incidence of complications occurring since implantation Revision rates and survival rates of prostheses

Study Groups Group 1: Subjects implanted with HUMELOCK I & II® Anatomic Shoulder System 2011 to 2013 Group 2: Subjects implanted with HUMELOCK II® Reversible System 2011 to 2013 Group 3: Subjects implanted with HUMELOCK Reversed® Shoulder System - 2012 - 2013 Group 4: Subjects implanted with EASYTECH® Anatomic Shoulder System - 2013 - 2014 Group 5: Subjects implanted with EASYTECH® Reversed Shoulder System (For Primary intention only) - 2013- 2014 Group 6: additional group for Subjects who were implanted with EASYTECH® Reversible Shoulder System (Exclusively for Revision of Easytech Anatomic) - 2013 -2014, if applicable Group 7: Subjects implanted with HUMERIS® Anatomic Shoulder System 2014 to 2015 Group 8: Subjects implanted with HUMERIS® Reversible Shoulder System 2014 to 2015

ELIGIBILITY:
Inclusion Criteria:

First of all, in order to be eligible to the study protocol, patients should have been treated primarily with one of studied device depending on surgeons' strategies' cares.

In order to be eligible to participate in this study, patients must meet all of the following criteria:

* Adult patient (≥ 18 years old) who received one of FX Solutions Shoulder System for indication of hemi or total shoulder replacement.
* Patient implanted between 2011 and 2015 with a minimum follow-up of 7 years
* Patient has been informed of his participation in a clinical study and did not object to data collection
* Patient insured with a social security system

Exclusion criteria for subject selection.

* Patient who does not meet the inclusion criteria above
* Protected adult
* People deprived of their liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Studied devices are intended for adult population that are treated for arthroplasty with the studied devices. These patients are presented a pathologic shoulder pain with origin with degeneration or trauma of the articulation pathologies.
  This study will include adult male and female patients from the Investigators' practice who were implanted with the FX Solution System; inclusion and exclusion criteria are defined not to introduce a too important bias of selection.
  The selected patients may be representative the overall population that could treated with devices.
Sampling Method: Non-Probability Sample
Enrollment: 416 (Estimated)
Dates: Start 2022-04-07 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Clinical outcomes | between 6 and 10 years depending on the date of implantation of the medical device in each treatment group
  Functional scores measurement with Constant-Murley's Score
Articular functional measurement scores | between 6 and 10 years depending on the date of implantation of the medical device in each treatment group
  measurement with American Shoulder and Elbow Surgeons Shoulder Score (ASES)
subjective evaluation by the patient of shoulder function | between 6 and 10 years depending on the date of implantation of the medical device in each treatment group
  Measurement with subjective shoulder value (SSV)

SECONDARY OUTCOMES:
Range of Motion scores | between 6 and 10 years depending on the date of implantation of the medical device in each treatment group
  Measurement of shoulder mobility (constant score)
Revision rate | between 6 and 10 years depending on the date of implantation of the medical device in each treatment group
  Number of patients with a change of implants out of the total number of patients reviewed in the study
Rate of complication | between 6 and 10 years depending on the date of implantation of the medical device in each treatment group
  All complications that had occurred will be collected in the CRF
Last information for patient lost to follow-up | between 6 and 10 years depending on the date of implantation of the medical device in each treatment group
  All available information about patients during his last medical follow-up
Survival rate | between 6 and 10 years depending on the date of implantation of the medical device in each treatment group
  Kaplan-Meier curve
Last information for deceased patient | between 6 and 10 years depending on the date of implantation of the medical device in each treatment group
  All available information about patients before his death

CONTACTS AND LOCATIONS:
Overall Officials: Laurent OBERT, MD, Principal Investigator — CHU Jean MINJOZ
Locations (20):
- France (19):
  - Hôpital Privé Antony, Antony
  - CHU Jean MINJOZ, Besançon
  - Centre hospitalier Bourg en Bresse, Bourg-en-Bresse
  - Clinique Convert, Bourg-en-Bresse
  - Infirmerie Protestante, Caluire-et-Cuire
  - Hopital privé Sainte Marie, Chalon-sur-Saône
  - CHMS Chambéry, Chambéry
  - Clinique La Montagne, Courbevoie
  - Centre Hospitalier de Dieppe, Dieppe
  - Clinique Bergouignan, Évreux
  - Clinique Saint Charles, Lyon
  - Clinique de l'Occitanie, Muret
  - Clinique Jouvenet, Paris
  - Clinique des Maussins, Paris
  - CHI Poissy - St Germain en Laye, Poissy
  - Hopital Privé Claude Gallien, Quincy-sous-Sénart
  - Clinique Mutualiste la Sagesse, Rennes
  - Centre Hospitalier de St Malo, St-Malo
  - Clinique Saint Léonard, Trélazé
- Centre Hospitalier Princesse Grace, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No
No plan to share IDP for this study

REFERENCES:
- [Background] Churchill RS. Stemless shoulder arthroplasty: current status. J Shoulder Elbow Surg. 2014 Sep;23(9):1409-14. doi: 10.1016/j.jse.2014.05.005. Epub 2014 Jul 11. PMID 25027481
- [Background] Cuff D, Pupello D, Virani N, Levy J, Frankle M. Reverse shoulder arthroplasty for the treatment of rotator cuff deficiency. J Bone Joint Surg Am. 2008 Jun;90(6):1244-51. doi: 10.2106/JBJS.G.00775. PMID 18519317
- [Background] De Wilde LF, Audenaert EA, Berghs BM. Shoulder prostheses treating cuff tear arthropathy: a comparative biomechanical study. J Orthop Res. 2004 Nov;22(6):1222-30. doi: 10.1016/j.orthres.2004.03.010. PMID 15475201
- [Background] Frankle M, Levy JC, Pupello D, Siegal S, Saleem A, Mighell M, Vasey M. The reverse shoulder prosthesis for glenohumeral arthritis associated with severe rotator cuff deficiency. a minimum two-year follow-up study of sixty patients surgical technique. J Bone Joint Surg Am. 2006 Sep;88 Suppl 1 Pt 2:178-90. doi: 10.2106/JBJS.F.00123. PMID 16951091
- [Background] Franklin JL, Barrett WP, Jackins SE, Matsen FA 3rd. Glenoid loosening in total shoulder arthroplasty. Association with rotator cuff deficiency. J Arthroplasty. 1988;3(1):39-46. doi: 10.1016/s0883-5403(88)80051-2. PMID 3361319
- [Background] Hawi N, Magosch P, Tauber M, Lichtenberg S, Habermeyer P. Nine-year outcome after anatomic stemless shoulder prosthesis: clinical and radiologic results. J Shoulder Elbow Surg. 2017 Sep;26(9):1609-1615. doi: 10.1016/j.jse.2017.02.017. Epub 2017 Apr 11. PMID 28410956
- [Background] Hawi N, Tauber M, Messina MJ, Habermeyer P, Martetschlager F. Anatomic stemless shoulder arthroplasty and related outcomes: a systematic review. BMC Musculoskelet Disord. 2016 Aug 30;17(1):376. doi: 10.1186/s12891-016-1235-0. PMID 27577859
- [Background] Jazayeri R, Kwon YW. Evolution of the reverse total shoulder prosthesis. Bull NYU Hosp Jt Dis. 2011;69(1):50-5. PMID 21332439
- [Background] Lugli T. Artificial shoulder joint by Pean (1893): the facts of an exceptional intervention and the prosthetic method. Clin Orthop Relat Res. 1978 Jun;(133):215-8. PMID 357063
- [Background] NEER CS 2nd. Articular replacement for the humeral head. J Bone Joint Surg Am. 1955 Apr;37-A(2):215-28. No abstract available. PMID 14367414
- [Background] Neer CS 2nd, Craig EV, Fukuda H. Cuff-tear arthropathy. J Bone Joint Surg Am. 1983 Dec;65(9):1232-44. PMID 6654936
- [Background] Neer CS 2nd, Watson KC, Stanton FJ. Recent experience in total shoulder replacement. J Bone Joint Surg Am. 1982 Mar;64(3):319-37. No abstract available. PMID 7061549
- [Background] Post M, Jablon M, Miller H, Singh M. Constrained total shoulder joint replacement: a critical review. Clin Orthop Relat Res. 1979 Oct;(144):135-50. PMID 535215